CLINICAL TRIAL: NCT00631176
Title: Effectiveness of "Just-In-Time" Training With/Without a High Fidelity Simulation on Patient Safety in Airway Management in Pediatric Intensive Care Unit
Brief Title: "Just-In-Time Training" in Pediatric Airway Management
Acronym: JIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Vinay Nadkarni, MD, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-8-4931; 5U18HS016678-02 (AHRQ)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Orotracheal Intubation
Keywords: oral intubation; just in time; simulation education; high fidelity training; intubation training; intubation success

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental)
  Interventions: Behavioral: Just-In-Time Training

INTERVENTIONS:
Behavioral: Just-In-Time Training — On-call pediatric residents from 7 south PICU (24 beds) will receive 20 minutes of just-in-time pediatric airway management training. This training will occur before their shift starts before the morning round. This training will cover direct laryngoscopy technique, orotracheal intubation technique, confirmation of the tube placement and recognition of associated events. This training will be done with or without high fidelity simulation function.
  Other Names: Over training; Intubation training; Rapid Refresher
  Arms: 2

SUMMARY:
This is a prospective interventional study to test the hypothesis that just-in-time training for pediatric airway management may improve patient safety and operational performance of orotracheal intubation and decreases intubation associated events in pediatric residents in the PICU. To test the hypothesis that high fidelity simulation may enhance the training efficacy and patient safety in simulation settings.

DETAILED DESCRIPTION:
Background:

Appropriate airway management is the most critical point in pediatric resuscitation and pediatric critical care. It remains, however, a challenge for pediatric residents to learn and retain this critical skill. Recent report from our PICU showed pediatric residents participated only 28% of initial orotracheal intubation, and the rate of the first successful endotracheal tube placement was only 38% of all orotracheal intubation attempt. Repetitive poor-skilled intubation attempts may be associated with complication such as dental or laryngeal contusion, and prolonged intubation attempt may be associated with hypoxia and hemodynamic instability. In order to improve the operational performance in the efficacy (first attempt success rate) and safety (minimizing the associated events which could potentially lead to adverse events), a better training method is warranted.

Objectives:

To test the hypothesis that just-in-time training for pediatric airway management may improve patient safety and operational performance of orotracheal intubation and decreases intubation associated events in pediatric residents in the PICU. To test the hypothesis that high fidelity simulation may enhance the training efficacy and patient safety in simulation settings.

Study Design:

This is a prospective interventional study. During the eighteen months of study period, one of two on-call pediatric residents from 7 south PICU (24 beds) will receive 20 minutes of just-in-time pediatric airway management training. This training will occur before their shift starts before the morning round. This training will cover direct laryngoscopy technique, orotracheal intubation technique, confirmation of the tube placement and recognition of associated events. This training will be done with or without high fidelity simulation function. We will use SimBaby (Laerdal, Norway). The assignment will be randomized. The clinical data of orotracheal intubation are collected through NEAR-4 KIDS registry. Primary outcome is a change in a first attempt success rate by the residents in an overtrained group (7 South PICU) compared to standard training group (7 East PICU). The secondary outcome is the rate of resident participation in orotracheal intubation attempt, the number of intubation attempt before successful intubation by residents and the number of intubation associated events. The videotaped performance during the training is analyzed with Healthcare Failure Mode and Effect Analysis (HFMEA) and will be compared between high fidelity simulation training group and low fidelity simulation training group. The evaluation system developed by HFMEA will be validated by a performance of experienced and non-experienced intubators. Furthermore, the real orotracheal intubation team performance in both PICUs will be evaluated with scale by a research assistant. The demographic and training data of participants of real PICU intubations will be collected. No patient identifiable information will be collected. This data will also be kept in a password-protected research computer.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric or Emergency Medicine Residents rotating through PICU in CHOP.

Exclusion Criteria:

1. Anesthesiology residents
2. Residents who had formal US training (ACGME accredited) in Neonatology or Pediatric Critical Care Medicine, Critical Care Medicine or Anesthesiology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the success of first intubation attempts by a resident. | per case

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Nadkarni, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States